CLINICAL TRIAL: NCT07116850
Title: Adjunctive Intermittent Theta-Burst Stimulation for First-Episode Schizophrenia: A Randomized Clinical Trial
Brief Title: Adjunctive iTBS for First-Episode Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Jiali Cui, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023S00450
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Disorder
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Adjunctive iTBS Group (Experimental): Participants (n=50) received risperidone (initiated at 1 mg/day and flexibly titrated to a maximum of 6 mg/day) and manualized Cognitive Behavioral Therapy (CBT) administered twice weekly for 12 weeks. In addition, they received active intermittent theta-burst stimulation (iTBS) for 20 sessions (5 days/week for 4 weeks) targeting the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Intermittent Theta-Burst Stimulation (iTBS); Drug: Risperidone; Behavioral: Cognitive Behavioral Therapy (CBT)
- Active Comparator: Control Group (Active Comparator): Participants (n=50) received an identical regimen of risperidone (initiated at 1 mg/day and flexibly titrated to a maximum of 6 mg/day) and manualized Cognitive Behavioral Therapy (CBT) administered twice weekly for 12 weeks, without iTBS.
  Interventions: Drug: Risperidone; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Device: Intermittent Theta-Burst Stimulation (iTBS) — Stimulation delivered using a Magstim RAPID2 stimulator. The target was the left DLPFC (F3 position). The protocol consisted of 20 sessions (5 days/week for 4 weeks) at 100% of the individual's motor threshold (MT), with each session delivering 2400 pulses.
  Arms: Experimental: Adjunctive iTBS Group
Drug: Risperidone — Oral risperidone (Jiangsu Enhua Pharmaceutical Co., Ltd.) initiated at 1 mg/day and flexibly titrated based on efficacy and tolerability to a maximum of 6 mg/day.
Behavioral: Cognitive Behavioral Therapy (CBT) — Manualized CBT administered twice weekly for 12 weeks. The therapy comprised an initial individual phase (4 weeks) focusing on psychoeducation and a subsequent group phase (8 weeks) targeting social and emotional skills.

SUMMARY:
This prospective, randomized, assessor-blinded study investigates the efficacy and safety of adding intermittent theta-burst stimulation (iTBS) to a standard treatment of risperidone and cognitive behavioral therapy (CBT) for patients with first-episode schizophrenia. The study aims to compare clinical symptom improvement, cognitive function changes, and levels of serum biomarkers (GDNF, CK-MB, DHEA-S) between a group receiving the combined therapy (iTBS+risperidone+CBT) and a control group receiving standard therapy (risperidone+CBT) over a 3-month period.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental disorder often treated with atypical antipsychotics like risperidone. However, pharmacotherapy alone has limited efficacy, especially for negative symptoms and cognitive deficits. Intermittent theta-burst stimulation (iTBS), a form of repetitive transcranial magnetic stimulation (rTMS), and cognitive behavioral therapy (CBT) are promising adjunctive treatments. This study was designed to prospectively evaluate the synergistic effects of a tripartite therapy. One hundred patients with first-episode schizophrenia were randomized to either an experimental group (iTBS + risperidone + CBT) or an active control group (risperidone + CBT). The primary objective was to assess the difference in clinical effective rate at 3 months, measured by the Positive and Negative Syndrome Scale (PANSS). Secondary objectives included evaluating changes in cognitive function (using subtests from the MATRICS Consensus Cognitive Battery), serum levels of potential biomarkers (GDNF, CK-MB, DHEA-S), and safety. The study aims to provide evidence for integrating iTBS into a multimodal treatment strategy for early-stage schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first-episode schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
* Age between 18 and 45 years.
* No prior antipsychotic treatment or a washout period of at least 4 weeks for any previous psychotropic medications.
* No contraindications to risperidone or iTBS.
* Educational level of junior high school or above, capable of understanding and completing study assessments.

Exclusion Criteria:

* Comorbid severe psychiatric disorders or significant organic brain disease.
* Pregnancy or lactation.
* Severe alcohol or substance dependence.
* Concurrent use of medications known to interact significantly with risperidone or affect cognitive function.
* Conditions that could interfere with cognitive assessment.
* Endocrine disorders, nutritional diseases, or epilepsy.
* History of cranial surgery or presence of metal implants in the head.
* Presence of biomedical devices (e.g., cardiac pacemakers).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total Effective Rate based on PANSS | 3 Months
  Clinical efficacy defined by the total effective rate based on the Positive and Negative Syndrome Scale (PANSS). The reduction rate is calculated as: (Baseline PANSS - Post-treatment PANSS) / (Baseline PANSS - 30). Total effective rate is the sum of participants achieving Cure (≥75% reduction), Marked Improvement (26%-74% reduction), or Effective (≥25% reduction).

SECONDARY OUTCOMES:
Change in Serum Glial Cell Line-Derived Neurotrophic Factor (GDNF) Level | Baseline, 3 Months
  Change in serum concentration of GDNF from baseline.
Change in Serum Creatine Kinase-MB (CK-MB) Level | Baseline, 3 Months
  Change in serum concentration of CK-MB from baseline.
Change in Serum Dehydroepiandrosterone Sulfate (DHEA-S) Level | Baseline, 3 Months
  Change in serum concentration of DHEA-S from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China